CLINICAL TRIAL: NCT00669591
Title: A Phase II Safety and Efficacy Study of Bavituximab Plus Docetaxel in Patients With Locally Advanced or Metastatic Breast Cancer
Brief Title: A Safety and Efficacy Study of Bavituximab Plus Docetaxel in Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPHM 0704
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: breast cancer; docetaxel chemotherapy; bavituximab; monoclonal antibody
MeSH Terms: conditions — Breast Neoplasms | interventions — bavituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients will receive up to six (6) 28-day cycles of docetaxel plus weekly bavituximab during the treatment phase. During the follow-up phase, patients will continue to receive weekly bavituximab until disease progression
  Interventions: Drug: Bavituximab

INTERVENTIONS:
Drug: Bavituximab — Weekly bavituximab infusion of 3 mg/kg combined with up to six 28-day cycles of docetaxel chemotherapy. After treatment phase, weekly bavituximab maintenance is continued until disease progression.

SUMMARY:
The purpose of the study is to determine the overall response to a combination of bavituximab and docetaxel in patients with advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Adult females over age 18 with life expectancy of at least 3 months
* Histologically or cytologically confirmed locally advanced or metastatic breast cancer
* One and only one prior chemotherapy regimen (no prior docetaxel)
* Measurable disease (at least one target lesion)at least 2 cm in longest diameter (1 cm by spiral CT)
* Adequate hematologic, renal, and hepatic function;

Exclusion Criteria:

* Known history of bleeding diathesis or coagulopathy
* Any current evidence of clinically significant bleeding
* Any history of thromboembolic events
* Concurrent hormone therapy
* Prior immunotherapy or radiotherapy to an area of measurable disease unless disease has recurred after radiotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete response + partial response) to a combination of bavituximab plus docetaxel in patients with metastatic breast cancer | Up to six (6) 28-day cycles of docetaxel plus weekly bavituximab until disease progression. After chemotherapy, weekly bavituximab is continued until disease progression. Approximate duration 1 year.

SECONDARY OUTCOMES:
Secondary objectives include time to tumor progression, duration of response, overall survival, and safety. | Approximately 1 year

CONTACTS AND LOCATIONS:
Locations (4):
- Georgia (4):
  - JSC. National Cancer Centre, Lisi Lake, K'alak'i T'bilisi
  - Ltd. Oncological Center, Batumi
  - Ltd. Tbilisi Oncological Dispensary, Tbilisi
  - Ltd. Chemotherapy and Immunotherapy clinic Medulla 6, Jikia Str, Tbilisi